CLINICAL TRIAL: NCT06465719
Title: A Multicenter, RAndomlzed, coNtrolled, umBrella Trial fOr Minimally Invasive Neurosurgery With Al-assisted Robotic Guidance for Moderate Basal Ganglia Hemorrhage (RAINBOW-MBH)
Brief Title: A Trial for Minimally Invasive Neurosurgery With AI-assisted Robotic Guidance for Moderate Basal Ganglia Hemorrhage (RAINBOW-MBH)
Acronym: RAINBOW-MBH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Huashan Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2024-0017
Record Dates: First submitted 2024-06-04; First posted 2024-06-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-08

CONDITIONS: Basal Ganglia Hemorrhage
MeSH Terms: conditions — Basal Ganglia Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients will be randomly assigned to treatment or conservative group, so masking is only for outcome assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tract-based AI Robot Guiding System Group (Experimental): Patients will be operated on minimally invasive puncture and aspiration using Tract-based AI Robot guidance System
  Interventions: Procedure: Minimally invasive basal ganglion hematoma evacuation with Tract-based AI Robot Guiding System
- Conservative Group (Sham Comparator): Patients will be managed with guideline-based medications without surgery
  Interventions: Drug: Patients will be managed with guideline-based medications

INTERVENTIONS:
Procedure: Minimally invasive basal ganglion hematoma evacuation with Tract-based AI Robot Guiding System — Basal ganglion hemorrhage patients will be operated on hematoma puncture and aspiration with Tract-based AI Robot Guiding System
  Other Names: Surgery Group
  Arms: Tract-based AI Robot Guiding System Group
Drug: Patients will be managed with guideline-based medications — Patients will be managed with guideline-based medications without surgery
  Other Names: Controlled Group
  Arms: Conservative Group

SUMMARY:
A nationwide, prospective, multicenter randomized controlled clinical trial to evaluate the therapeutic effects of the fiber tract-based artificial intelligence (AI) Robot Guiding System on the perioperative and long-term recovery of patients with moderate-volume basal ganglion hemorrhage.

DETAILED DESCRIPTION:
Basal ganglion hemorrhage is one of the most common subtypes of cerebral hemorrhage, characterized by high morbidity, mortality, and disability rates. Minimally invasive surgery for cerebral hemorrhage, particularly utilizing a fiber tract-based AI Robot Guiding System, has shown potential advantages for patient prognosis. However, there is currently no standardized practice or robust evidence confirming the effectiveness and safety of this technology for small-volume basal ganglion hemorrhage. Therefore, we are conducting a nationwide, prospective, multicenter randomized controlled clinical trial to evaluate the therapeutic effects of the fiber tract-based artificial intelligence (AI) Robot Guiding System on the perioperative and long-term recovery of patients with moderate-volume basal ganglion hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at randomization
2. Hypertensive basal ganglia hemorrhage confirmed by CT/CTA
3. Hematoma volume 15-30 mL (excluding 30 mL)
4. Functional impairment (aphasia, hemiparesis with strength ≤3, or NIHSS ≥15)
5. CT shows stable hematoma (≥6h interval, change <5 mL)
6. GCS ≥9
7. Surgery feasible within 72h after onset
8. Pre-ICH mRS ≤1
9. Informed consent obtained according to laws and ethics

Exclusion Criteria:

1. Hematoma involving the thalamus, midbrain, or other areas
2. Radiologically diagnosed cerebrovascular abnormalities, as well as ischemic infarction converting to intracerebral hemorrhage, or recent (within 1 year) recurrence of intracerebral hemorrhage
3. Signs of impending brain herniation, such as midline shift >1 cm or changes in the ipsilateral pupil;
4. Any irreversible coagulopathy disorders or known coagulation system disease; platelet count <100,000; INR >1.4; use of anticoagulants within 7 days prior to this hemorrhage;
5. Pregnant or possibly pregnant
6. Patients with severe concomitant diseases that may interfere with outcome assessment
7. Poor compliance or follow-up difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Utility-weighted modified Rankin Scale (UW-mRS) | 6 months
  The mRS is a 7-level ordinal scale used to evaluate functional outcomes after stroke. The categories are defined as follows:
  0 = No symptoms；
  1. = No significant disability. Able to carry out all usual activities, despite some symptoms；
  2. = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities；
  3. = Moderate disability. Requires some help, but able to walk unassisted；
  4. = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted；
  5. = Severe disability. Requires constant nursing care and attention, bedridden, incontinent；
  6. = Dead； Utility-weighted modified Rankin Scale (UW-mRS), which applies utility values to each mRS category as shown below： mRS 0= UW-mRS 1；mRS 1= UW-mRS 0.91; mRS 2= UW-mRS 0.76; mRS 3= UW-mRS 0.65; mRS 4= UW-mRS 0.33; mRS 5= UW-mRS 0; mRS 6= UW-mRS 0.

SECONDARY OUTCOMES:
Ordinal shift in modified Rankin Scale | 6 months
  Ordinal shift analysis of the modified Rankin Scale (mRS), which measures the degree of disability or dependence in daily activities after stroke. The scale ranges from 0 (no symptoms) to 6 (death). This outcome assesses whether there is a shift toward better or worse functional status across the full ordinal distribution of mRS scores.
Excellent functional neurological outcome | 6 months
  Excellent functional neurological outcome means modified Rankin scale (mRS) scores 0-1. The minimum mRS is 0 (no symptoms) while the maximum mRS is 6 (death). The higher the mRS score is the worse outcome is.
Independent functional neurological outcome | 6 months
  Independent functional neurological outcome means modified Rankin scale (mRS) scores 0-2. The minimum mRS is 0 (no symptoms) while the maximum mRS is 6 (death). The higher the mRS score is the worse outcome is.
Health Related Quality of Life | 6 months
  Health Related Quality of Life based on EuroQol 5 Dimension 5 Level (EQ-5D-5L).The EQ-5D-5L is a generic instrument for describing and valuing health. It assesses five domains: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has five response categories corresponding to: no problems, slight, moderate, severe and extreme problems.
Total length of hospital stay | 6 months
  Total length of hospital stay refers to the number of days from the date of hospital admission to the date of discharge.
AD8 Dementia Screening | 6 months
  The AD8 (Eight-item Interview to Differentiate Aging and Dementia) is a brief screening tool designed to distinguish normal aging from possible dementia. The AD8 focuses on changes in memory, orientation, judgment, and daily activities. A greater number of "Yes" responses indicates higher likelihood of cognitive impairment or dementia, warranting further diagnostic evaluation.
Hematoma evacuation rate | 30 days after treatment
  Hematoma clearance rate at Day1 and Day30 after treatment
Total medical expenses during hospitalization | 6 month
  Total medical expenses during hospitalization

OTHER OUTCOMES:
Mortality | 6 months
  Mortality status equals to death which will be collected at all visits during the trial period
Serious Adverse Events (SAEs) | 6 months
  The reporting and notification of SAEs follows ICH-GCP guidelines. According to the WHO International Drug Monitoring Centre (1994), an SAE is any adverse medical event that: Leading to death; Life-threatening; Requires hospitalization or prolongs existing hospitalization; Results in persistent or significant disability/incapacity; Congenital anomaly/birth defect; etc.

CONTACTS AND LOCATIONS:
Overall Officials: Gao Chen, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Multicenter, Randomized, Controlled, Umbrella Trial for Minimally Invasive Neurosurgery With Al-assisted Robotic Guidance for Hemorrhagic Stroke (RAINBOW-ICH) — https://clinicaltrials.gov/study/NCT07205263